CLINICAL TRIAL: NCT07197697
Title: A Phase II Exploratory Study of Iparomlimab and Tuvonralimab Combined With Chemotherapy in Neoadjuvant Treatment of HR+/HER2- Breast Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yue-Yin Pan, chief physicians, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-LLYJ-0007
Record Dates: First submitted 2025-09-02; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Iparomlimab and Tuvonralimab combined with chemotherapy
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection (QL1706) combined chemotherapy

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection (QL1706) combined chemotherapy — The dosage of Iparomlimab and Tuvonralimab Injection is 5mg/kg, administered intravenously, with each treatment cycle lasting every 3 weeks. The chemotherapy regimen is AC-T: epirubicin 100mg/m2, cyclophosphamide 600mg/m2, every 3 weeks for 4 cycles; followed by paclitaxel 80mg/m2, every week for 12 cycles. A total of 8 cycles of neoadjuvant chemotherapy combined with immunotherapy were performed before the surgery. It is recommended that the surgery be conducted within 4 weeks after the completion of neoadjuvant treatment. The postoperative adjuvant treatment can be continued with postoperative adjuvant chemotherapy and the treatment of the etolo combination antibody according to the decision of the researcher and/or the willingness of the subject.

SUMMARY:
This study is a prospective, multicenter, single-arm, exploratory study. 30 patients with locally advanced HR+/HER2- breast cancer who have not received any treatment were recruited to receive apalutamide voraparib combined with chemotherapy for neoadjuvant therapy. This study adopts Simon's two-stage design: in the first stage, 12 patients need to be enrolled. If among these 12 patients, 1 or fewer patients achieve tpCR, the study will be prematurely terminated due to early failure. Otherwise, 18 patients will be enrolled in the second stage. If 7 or more patients achieve tpCR among the 30 patients, the study achieves the expected results, and the drug can be further studied; otherwise, the study fails, and the drug does not need further study. The aim of this study is to evaluate the efficacy and safety of apalutamide voraparib combined with chemotherapy for neoadjuvant therapy in patients with HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient must meet all of the following criteria to be included in the study:

  1. Age ≥ 18 years and ≤ 75 years, regardless of gender;
  2. The primary lesion tissue pathology is confirmed as HR+/HER2- breast cancer, following the 2018 ASCO/CAP breast cancer HER2 testing guidelines and the 2010 ASCO/CAP breast cancer ER/PR testing guidelines for interpretation. HER2-negative is defined as confirmed by the pathology laboratory with an immunohistochemistry (IHC) score of HER2 0/1+ or 2+ and negative in in situ hybridization (ISH), and estrogen receptor positive (ER+) breast cancer with or without progesterone receptor (PgR) expression;
  3. Tumor histological grade 3, or histological grade 2 with the percentage of ER expression level between 1-10%;
  4. According to the American Joint Committee on Cancer (AJCC) 8th edition TNM classification, the clinical stage should be T1c-T2cN1-2 or T3-4cN0-2, M0 stage;
  5. At least one measurable lesion (in accordance with the RECIST 1.1 version standard);
  6. Expected survival time ≥ 12 weeks;
  7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
  8. The subject has no severe blood, heart, lung, liver, or kidney function abnormalities and immunodeficiency diseases. The functional level of important organs within one week before the first administration must meet the following requirements:

     1. Blood routine: HGB ≥ 90g/L; WBC ≥ 4.0×109/L; NEUT ≥ 2.0×109/L; PLT ≥ 100×109/L;
     2. Blood biochemistry: TBIL ≤ 1.5×ULN; ALT and AST ≤ 3×ULN (for those with liver metastasis, ALT and AST ≤ 5×ULN); BUN and Cr ≤ 1.5×ULN and creatinine clearance rate ≥ 50 mL/min;
     3. Cardiac color Doppler ultrasound before the first administration must meet: left ventricular ejection fraction (LVEF) > 50%;
  9. Thyroid stimulating hormone (TSH) ≤ upper limit of normal (ULN); if abnormal, T3 and T4 levels should be examined; if T3 and T4 levels are normal, the subject can be included;
  10. Pregnant patients should have a negative pregnancy test and voluntarily take effective and reliable contraceptive measures during the test period;
  11. The subject voluntarily joins this study, signs the informed consent, has good compliance and is willing to cooperate with follow-up.

Exclusion Criteria:

* If the patient meets any of the following conditions, they will not be eligible:

  1. Patients with stage IV metastatic breast cancer or other conditions deemed by the researchers as not achievable through neoadjuvant therapy for radical surgical resection;
  2. Bilateral invasive breast cancer;
  3. Breast cancer patients who have previously received anti-tumor treatments such as chemotherapy, endocrine therapy, or undergone breast surgery (except for the diagnostic biopsy of primary breast cancer);
  4. Patients who participated in other drug clinical trials within 4 weeks prior to enrollment, received major surgical treatment, incisional biopsy, or significant traumatic injury (except for the diagnostic biopsy of primary breast cancer);
  5. Within 4 weeks before the first administration or planned to receive attenuated live vaccines during the study;
  6. Patients with other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or papillary thyroid carcinoma;
  7. Patients receiving any other anti-tumor treatment simultaneously;
  8. Patients with a known history of allergy to the components of this study drug;
  9. Patients with a clear history of neurological or mental disorders, including epilepsy or dementia, or a history of substance abuse or drug use for mental disorders;
  10. Patients with a known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
  11. Pregnant or lactating female patients, or female patients with reproductive capacity and positive baseline pregnancy test results;
  12. Patients with active infectious diseases;
  13. Diagnosed with immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy;
  14. Patients with active or potentially recurrent autoimmune diseases, except for: vitiligo, alopecia, psoriasis or eczema that do not require systemic treatment; hypothyroidism caused by autoimmune thyroiditis, requiring only a stable dose of hormone replacement therapy; type 1 diabetes requiring only a stable dose of insulin replacement therapy;
  15. According to the investigator's judgment, there are serious diseases that endanger the patient's safety or affect the patient's ability to complete the study (including but not limited to drug-controlled interstitial lung disease, severe pulmonary dysfunction/disease, cerebrovascular accident, severe diabetes);
  16. Excluded patients with any of the following cardiovascular diseases:

      1. Within 6 months before the first administration, experienced myocardial infarction, unstable angina pectoris, pulmonary embolism, acute/ persistent myocardial ischemia, cerebrovascular accident, transient cerebral ischemic attack, or other clinically significant/ requiring drug treatment intervention thromboembolic or ischemic events;
      2. Had NYHA III-IV grade congestive heart failure in the past and/or currently;
      3. Had severe arrhythmias that require drug treatment in the past and/or currently;
      4. Within 12-lead ECG before the first administration showed a mean QT interval (QTcF) > 470 ms.
  17. The investigator determines that the patient is not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
tpCR rate，total physiological complex response | From the time of enrollment to one month after the surgery
  After the resection of the primary tumor, microscopic examination of the breast and the ipsilateral axillary lymph nodes revealed no invasive tumor cells (ypT0/is ypN0)

SECONDARY OUTCOMES:
bpCR，breast physiological complex response | From the time of enrollment to one month after the surgery
  After the primary tumor was removed, microscopic examination of the breast revealed no invasive tumor cells (ypT0/is)
EFS，Event-free survival | baseline，1year，up to 2year
  The time from the start of medication to the occurrence of any of the following events for the first time: disease progression making surgical treatment impossible, local or distant recurrence, death due to any cause, etc.
ORR，Objective Response Rate | 6-12 months
  The proportion of patients whose tumor volume has decreased by 30% and has remained stable for more than four weeks is referred to as the sum of complete response (CR) and partial response (PR).
OS，Overall Survival | baseline，1year，up to 2year
  Refers to the period from the start of medication use until death occurs due to any cause.
adverse event | up to 2year
  Collect all adverse events that occurred in all subjects from the signing of the informed consent to 28 days after the cessation of medication, including clinical symptoms and abnormal vital signs, as well as abnormalities in laboratory tests. Record the clinical manifestations, severity, occurrence time, duration, treatment methods, prognosis, and determine the correlation between these events and the test drug.
PRO | through study completion, an average of 1 year
  Outcome indicators reported by the patients，Score using the Chinese version of the EORTC Quality of Life Questionnaire Core 30 (QLQ-C30, V3.0)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol